CLINICAL TRIAL: NCT02449187
Title: A Randomized, Open-label, Single Dose, Crossover Study to Investigate the Effect of Food on the Pharmacokinetics of JLP-1310 in Healthy Male Volunteers
Brief Title: Investigate the Effect of Food on the Pharmacokinetics of JLP-1310 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1310-102-FE
Record Dates: First submitted 2015-05-13; First posted 2015-05-20 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Diabetes; Hyperlipidemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias | interventions — Metformin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JLP-1310, Fasted followed by fed (Experimental): JLP-1310 dosing in the fasted state followed by fed dosing
  Interventions:
  Drug: JLP-1310
  Interventions: Drug: JLP-1310, Fasted followed by fed
- JLP-1310, Fed followed by fasted (Experimental): JLP-1310 dosing in the fasted state followed by fed dosing
  Interventions:
  Drug: JLP-1310
  Interventions: Drug: JLP-1310, Fed followed by fasted

INTERVENTIONS:
Drug: JLP-1310, Fasted followed by fed — In period 1, the subjects will receive an oral pill of JLP-1310 under fasted condition.
  In period 2, the subjects will receive an oral pill of JLP-1310 under fed condition.
  Other Names: metformin hydrochloride, rosuvastatin calcium
  Arms: JLP-1310, Fasted followed by fed
Drug: JLP-1310, Fed followed by fasted — In period 1, the subjects will receive an oral pill of JLP-1310 under fed condition.
  In period 2, the subjects will receive an oral pill of JLP-1310 under fasted condition.
  Other Names: metformin hydrochloride, rosuvastatin calcium
  Arms: JLP-1310, Fed followed by fasted

SUMMARY:
A randomized, open-label, single dose, crossover study to investigate the effect of food on the pharmacokinetics of JLP-1310 in healthy male volunteers.

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer, age is over 19 years
2. Body weight is over 55kg, The result of Body Mass Index(BMI) is not less than 17.5 kg/m2 , no more than 30.5 kg/m2
3. Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial
4. Subject who has the ability and willingness to participate the whole period of trial

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Subjects who are allergic to investigational drug.
3. Subjects who have a medical history which can affect the clinical trial.
4. Hypertension(Systolic BP ≥ 140mmHG or Diastolic BP ≥ 90mmHg), Liver enzyme (AST, ALT) level exceeds the maximum normal range more than one and a half times.
5. History of drug abuse or positive drug screening.
6. Participation in other drug studies within 3 months prior to the drug administration.
7. Whole blood donation within 60 days, blood component donation within 30 days or who got transfusion within 30days.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Cmax | 48 hours from baseline
AUC(last) | 48 hours from baseline

SECONDARY OUTCOMES:
AUC(inf) | 48 hours from baseline
Tmax | 48 hours from baseline
T1/2 | 48 hours from baseline
CL/F | 48 hours from baseline
Vd/F | 48 hours from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sang Heon Cho, MD., Ph.D, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No